CLINICAL TRIAL: NCT02812589
Title: Improving the Specificity of Breast MRI Through Diffusion Tensor Breast MRI (DTI)
Brief Title: Diffusion Tensor Breast MRI (DTI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-6856-CE
Record Dates: First submitted 2016-05-04; First posted 2016-06-24 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diffusion tensor imaging (DTI) in breast MRI (Experimental)
  Interventions: Other: Diffusion tensor imaging (DTI) in Breast MRI

INTERVENTIONS:
Other: Diffusion tensor imaging (DTI) in Breast MRI

SUMMARY:
The breast MRI is used in the preoperative scenario to evaluate the extension of a newly diagnosed breast cancer and to screen the contralateral breast. The scan consists of a series of images taken after the use of intravascular contrast media that may detect areas of enhancement that look malignant, but are actually benign tissue, producing a false positive result. The investigators aim to evaluate a novel MRI sequence of images that does not use contrast, diffusion tensor imaging (DTI). Addition of DTI sequence does not add significantly to the time of standard breast MRI exam. This novel technique provides improved detection of tissue microstructure and is able to differentiate malignant from benign tumor. Hence, the investigators hypothesize that DTI may decrease the false positive rate when compared with standard dynamic contrast-enhanced (DCE) MRI.

ELIGIBILITY:
Inclusion Criteria:

* Female of any race, ethnicity and lifetime risk.
* Eighteen years or older.
* Known recent diagnosis of a breast cancer and normal clinical breast exam of the contralateral side.
* Self-detected lump suspicious for breast cancer that it has not been biopsied yet.

Exclusion Criteria:

* Inability to understand the consent form
* Pregnant or nursing
* Currently taking tamoxifen, evista (raloxifene), or an aromatase inhibitor for adjuvant therapy or chemoprevention
* Physically unable to lie down on her belly for at least 10 minutes.
* Have had benign needle biopsy of the breast performed within 3 months, or breast surgery within 1 year prior to MRI exam.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Validate DTI as a valuable adjunct to improve lesion characterization on breast MRI by using the difference in recall rates | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anabel Scaranelo, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, University Health Network, 610 University Ave., Toronto, Ontario, Canada